CLINICAL TRIAL: NCT05931120
Title: Comparative Effects of Dry Needling and Instrument Assisted Soft Tissue Mobilization on Hamstring Tightness in Patients With Posterior Pelvic Tilt.
Brief Title: Comparison of Dry Needling and IASTM on Hamstring Tightness in Posterior Pelvic Tilt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0149
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hamstring Contractures
Keywords: dry needling; Hamstring tightness; IASTM; Posterior pelvic tilt
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): dry needling with multimodal physical therapy approach containing hurdler stretch and extended triangular pose
  Interventions: Device: Dry needling
- IASTM (Experimental): IASTM with multimodal physical therapy approach containing hurdler stretch and extended triangular pose
  Interventions: Device: IASTM

INTERVENTIONS:
Device: Dry needling — dry needling using 50mm or 60mm sized needles based on individual muscle bulk. Targeted dry needling will be performed on the muscles presenting with tight hamstrings. hurdler Hamstring stretch, extended triangular pose 10 repetitions, 3 sets per session and 2 sessions per week for 4weeks.
  total 8 sessions , each consisting of 40mins
  Arms: Dry needling
Device: IASTM — Instrument assisted soft tissue mobilization tools targeting tight hamstrings. hurdler Hamstring stretch, extended triangular pose 10 repetitions, 3 sets per session and 2 sessions per week for 4weeks.
  total 8 sessions , each consisting of 40mins
  Arms: IASTM

SUMMARY:
The purpose of the study is to compare the effects of dry needling (DN) and instrument-assisted soft tissue mobilization (IASTM) on pain, range of motion, lower extremity functional status on hamstring tightness in patients with posterior pelvic tilt.

DETAILED DESCRIPTION:
A study conducted analyzed the effects of a 3-week combined treatment using transcutaneous electrical nerve stimulation (TENS) and instrument-assisted soft tissue mobilization (IASTM) on chronic back pain. The findings showed that this short-term combined treatment led to reduced pain levels and improved motor function in Chronic low back pain (CLBP) patients. These results suggest that TENS and IASTM could be beneficial as a complementary approach for managing chronic low back pain.

In a randomized trial which shows the results by comparing the efficacy of dry needling (DN) and Graston techniques (GR) in treating upper trapezius myofascial trigger points. Both interventions, were administered twice a week for 2 weeks and when combined with conventional treatment and home exercises, showed significant improvements. However, DN demonstrated superior outcomes in terms of the myofascial diagnostic scale, neck disability index, pain rating, and cervical range of motion. These findings highlight the effectiveness of DN in targeting trigger points and optimizing clinical outcomes.

A notable lacuna persists in the literature concerning the effects of dry needling (DN) and instrument-assisted soft tissue mobilization (IASTM) on patients diagnosed with hamstring tightness and concurrent posterior pelvic tilt. The dearth of comparative research, inadequate incorporation of comprehensive outcome measures, and the paucity of studies targeting this specific patient cohort contribute to this research gap. Addressing this gap would yield valuable insights into the comparative efficacies and outcomes of DN and IASTM pertaining to pain modulation, range of motion enhancement and optimization of lower extremity functional status in this distinct population subset.

ELIGIBILITY:
Inclusion Criteria:

* Lack of greater or equal to 20 degrees of supine active knee extension
* Passive SLR less or equal to 75 degrees
* Atraumatic back or knee pain greater or equal to 2 weeks
* Individuals willing to participate in the required treatment sessions and follow-up assessments
* Posterior pelvic tilt 8.9 standard deviation of 4.5 degree

Exclusion Criteria:

* History of herniated lumbar disc/radiculopathy
* Prior surgery in the hip, knee, or back
* Self-reported pregnancy
* History of blood borne pathogens/infectious disease/active infection
* Metal allergy
* Positive instability tests indicative of ligamentous tear
* Positive meniscal tests

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-02-08 (Estimated)

PRIMARY OUTCOMES:
ROM( Posterior pelvic tilt) | 4th week
  The pelvic tilt is the angle between the horizontal plan and a line drawn from the anterior superior iliac spine (ASIS) to the posterior superior iliac spine (PSIS) in quiet standing. The average ranges of anterior and posterior pelvic tilting are 13.0 ± 4.9°, and 8.9 ± 4.5°,
ROM(AKE) | 4th week
  The Active Knee Extension Test is used to assess hamstring muscle length and the range of active knee extension in the position of hip flexion.The subject is positioned on the examination table in supine, the lower limb that is'nt examined is positioned in stabilised on the support surface. The opposite limb is elevated so that the hip is in 90degrees of flexion and the knees are extended to reach a position perpendicular to the ground. A lag of 20degrees is considered normal from full extension, anything less than 20degrees is considered as hamstrings tightness. This range needs to be measure using a digital inclinometer
ROM(SLR) | 4th week
  The straight leg raise or straight leg lift is a hamstring muscle flexibility test. While the subject is lying on their back, the straight leg is raised as far as possible, and the angle of the leg from the horizontal is measured.
  The straight leg raise test measures hamstring tightness. Restricted flexibility in the hamstrings will contribute to lower back, pelvis, hip, and knee malalignment. The straight leg raise test focuses on proximal hamstring tightness. The test is performed passively.

SECONDARY OUTCOMES:
Numeric pain rating scale | 4th week
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

OTHER OUTCOMES:
lower extremity functional scale | 4th week
  The lower extremity functional scale (LEFS) is a valid patient-rated outcome measure (PROM) for the measurement of lower extremity function.
  The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, phD, Principal Investigator — Riphah International University
Locations (1):
- DHQ Nankana sahib, Nankana Sahib, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allam NM, Eladl HM, Elruwaili LT, Elruwaili LF, Elbenya TJ, Elanzi EM, Elquobisi FF, Elgadoa HM, Elghaleb MA, Elsaeid MS, Elquarenes RA, Elrashed SM, Elmobarak SS, Elkholi SM, Eid MM, Alanazi AM, Nambi G, Abdelbasset WK. Correlation between hamstring muscle tightness and incidence of low back pain in female students at Jouf University, Saudi Arabia. Eur Rev Med Pharmacol Sci. 2022 Nov;26(21):7779-7787. doi: 10.26355/eurrev_202211_30127. PMID 36394725
- [Background] Dhingani M, Mody V. Short Term Effects of Remote Myofascial Release versus Mulligan's Bent Leg Raise on Hamstring and Lumbar Spine Flexibility in College Going Students: An Experimental Study. Indian Journal of Physiotherapy & Occupational Therapy Print-(ISSN 0973-5666) and Electronic-(ISSN 0973-5674). 2022;16(2):106-13.
- [Background] Suhail M, Prakash A, Sonali D, Sangeeta M. Effectiveness of dynamic soft tissue mobilization vs passive stretching to improve hamstring flexibility in stroke patients-A comparative study. 2022.
- [Background] Raza A, Haq K, Naveed J, Ali S, Rizwan I. Immediate effects of post facilitation stretch technique on straight leg raise with/without thoraco-lumber direct myofacial release in non-symptomatic adults. The Rehabilitation Journal. 2022;6(04):462-7.
- [Background] Sathe SS, Rajandekar T, Thodge K, Gawande V. Comparison between immediate effects of MET and passive stretching techniques on hamstring flexibility in patients with hamstring tightness: An experimental study. Indian Journal of Forensic Medicine & Toxicology. 2020;14(4):6857-62.
- [Background] Ansari NN, Alaei P, Naghdi S, Fakhari Z, Komesh S, Dommerholt J. Immediate Effects of Dry Needling as a Novel Strategy for Hamstring Flexibility: A Single-Blinded Clinical Pilot Study. J Sport Rehabil. 2020 Feb 1;29(2):156-161. doi: 10.1123/jsr.2018-0013. PMID 30526283
- [Background] Noreen A, Rashad A, Naeem F, Intikhab R, Angela C, Sonia A, et al. Comparative effect of graston technique and muscle energy technique on the flexibility of hamstring muscle. International Journal of Clinical Skills. 2022;16(8):255.
- [Background] Clark NG. The Neurophysiological Effects of Dry Needling to the Thoracolumbar Junction Multifidi in Subjects with Low Back Pain and Decreased Hamstring Length: Nova Southeastern University; 2020.
- [Background] Kim YK, Cho SY, Lee KH. Effects of transcutaneous electrical nerve stimulation and instrument-assisted soft tissue mobilization combined treatment on chronic low back pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2021;34(5):895-902. doi: 10.3233/BMR-200369. PMID 34092603
- [Background] Vicente-Mampel J, Bautista IJ, Lopez-Soler J, Torregrosa-Valls J, Falaguera-Vera F, Gargallo P, Baraja-Vegas L. Acute effects of self-myofascial release compared to dry needling on myofascial pain syndrome related outcomes: Range of motion, muscle soreness and performance. A randomized controlled trial. J Bodyw Mov Ther. 2024 Oct;40:632-639. doi: 10.1016/j.jbmt.2024.04.005. Epub 2024 Apr 10. PMID 39593656
- [Background] Osailan A, Jamaan A, Talha K, Alhndi M. Instrument assisted soft tissue mobilization (IASTM) versus stretching: A comparison in effectiveness on hip active range of motion, muscle torque and power in people with hamstring tightness. J Bodyw Mov Ther. 2021 Jul;27:200-206. doi: 10.1016/j.jbmt.2021.03.001. Epub 2021 Mar 11. PMID 34391234
- [Background] 羅佳安. The Effects of Dry Needling on Gait Patterns in Subjects with Hamstring Muscle Fatigue 2021.
- [Background] Sanchez-Infante J, Navarro-Santana MJ, Bravo-Sanchez A, Jimenez-Diaz F, Abian-Vicen J. Is Dry Needling Applied by Physical Therapists Effective for Pain in Musculoskeletal Conditions? A Systematic Review and Meta-Analysis. Phys Ther. 2021 Mar 3;101(3):pzab070. doi: 10.1093/ptj/pzab070. PMID 33609356
- [Background] Haq K, Riaz H. Comparison of dry needling and Graston technique on Active Myofascial trigger points in upper trapezius. Rawal Medical Journal. 2022;47(1):129-.
- [Background] Chintamani R, Metgud S, Heggannavar A. Short term effects of instrument assisted soft tissuemobilisation technique versus Mulligan's bent leg raise technique in asymptomatic subjects with hamstring tightness-a randomised clinical trial. Int J Health Sci Res. 2019;9:50-64.
- [Background] Kamble S, Chintamani R, Jagtap V. Short Term Effect of Isolytic Contraction on Hamstring Flexibility in Asymptomatic Subjects with Hamstring Tightness: A Randomised Controlled Trial. Indian Journal of Public Health Research & Development. 2020;11(2).
- [Background] Putra DP, Sari GM, Utomo DN. Different Effect of Static Stretching and Neurodynamic Technique in Increasing Hamstring Flexibility on Hamstring Tightness. Different Effect of Static Stretching and Neurodynamic Technique in Increasing Hamstring Flexibility on Hamstring Tightness. 2021;86(1):6-.
- [Background] Kim J, Kim H, Lee J, Lee H, Jung H, Cho Y, et al. Changes in the quadriceps-to-hamstring muscle ratio during wall squatting according to the straight leg raise test angle. Physical Therapy Rehabilitation Science. 2019;8(1):45-51.
- [Background] Sadat A, Otadi K, Fakhari Z, Nakhostin Ansari N, Bagheri H, Ghorbanpour A. The effects of dry needling on flexibility & electrophysiological indices in healthy men with hamstring tightness: double-blind, randomized, placebo-controlled trial. Tehran University Medical Journal TUMS Publications. 2020;78(7):442-7.
- [Background] Shaikh SM, Moharkar AC. Effect of core stability exercises versus Surya Namaskar on hamstring tightness in healthy adults using active knee extension test at the end of 6 weeks: A comparative study. IJAR. 2020;6(3):386-90.
- [Background] Deshpande K, Dhumale S. Effect of muscle energy technique v/s static stretching on tight hamstring muscles length and pelvic inclination amongst asymptomatic adults
- [Background] Doeringer JR, Ramirez R, Colas M. Instrument-Assisted Soft Tissue Mobilization Increased Hamstring Mobility. J Sport Rehabil. 2022 Aug 11;32(2):165-169. doi: 10.1123/jsr.2022-0015. Print 2023 Feb 1. PMID 35961647
- [Background] Naweed J, Razzaq M, Sheraz S, Anwar N, Sadiq N, Naweed S. Comparison of active isolated stretch and post isometric relaxation for improving hamstring flexibility in young healthy adults. Pakistan Armed Forces Medical Journal. 2020;70(3):770-75.